CLINICAL TRIAL: NCT00584714
Title: Long-Term Follow-Up of Selected Patients Enrolled in Phase 3 Clinical Trial 127-014 Using PB127 Ultrasound Imaging Agent
Brief Title: Long-Term Follow-up Study of Patients Who Received PB127 Ultrasound Imaging Agent
Status: Terminated | Type: Observational
Why Stopped: Discontinued PB127 development program for business reasons
Sponsor: Point Biomedical (Industry)
Responsible Party: Tom Ottoboni PhD/Chief Operating Officer, POINT Biomedical Corp.
Other Study IDs: 127-014-A
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: Coronary Artery Disease
Keywords: ultrasound; perfusion; SPECT; coronary artery disease; chest pain; low probability; angiography; clinical outcomes
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect longer term follow-up information concerning health and survival on selected patients who received PB127 for injectable suspension in the pivotal trial (127-014).

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in Protocol 127-014 who

1. Were enrolled in Stratum 1
2. Did not undergo angiography during study evaluation
3. Did not have a clinical oucome during the initial 6 month follow-up period as described in Protocol 127-014.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with low/very low pre-test probability of coronary artery disease enrolled in Protocol 127-014 who did not have or were not schedule to undergo coronary angiography at the time of enrollment and did not have a clinical outcome during the initial 6 month follow-up period.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To collect longer-term follow-up clinical information on selected patients enrolled in Protocol 127-014 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ehlgen, MD, PhD, Study Director — POINT Biomedical Corp.
Locations (39):
- United States (39):
  - University of Arizona Saver Heart Clinic, Tucson, Arizona
  - Cardiovascular Associates of the Peninsula, Burlingame, California
  - Long Beach VA Medical Center Cardiology Division, Long Beach, California
  - Cedars Sinai Medical Center Division of Cardiology, Los Angeles, California
  - Sutter Roseville Medical Center, Roseville, California
  - University of California San Diego Division of Cardiology, San Diego, California
  - San Francisco VA Medical Center NCIRE, San Francisco, California
  - Connecticut Clinical Research, Bridgeport, Connecticut
  - Alfieri Cardiology, Newark, Delaware
  - Washington Hospital Center Cardiovascular Research Institute, Washington D.C., District of Columbia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Midwest Cardiology Associates, Overland Park, Kansas
  - The Center for Cardiovascular Studies Kramer & Crouse Cardiology, Shawnee Mission, Kansas
  - Western Baptist Hospital The Heart Group, Paducah, Kentucky
  - Androscoggin Cardiovascular Associates, Auburn, Maine
  - Maine Cardiology Associates, South Portland, Maine
  - Brigham & Women's Hosptial, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Department of Cardiology, Rochester, Minnesota
  - Cardiovascular Consultants, Kansas City, Missouri
  - St. Louis University Medical Center, St Louis, Missouri
  - North Shore University Hospital, Manhasset, New York
  - St. Luke's Roosevelt Hospital Echocardiography Lab, New York, New York
  - Stonybrook University Medical Center, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Carolina Cardiology Associates, High Point, North Carolina
  - The Cleveland Clinic Foundation Department of Cardiology, Cleveland, Ohio
  - Ohio State University College of Medicine and Public Health, Columbus, Ohio
  - University of Pittsburgh Cardiovascular Institute, Pittsburgh, Pennsylvania
  - Seton Healthcare Network Brackenridge Hospital, Austin, Texas
  - Austin Heart, Austin, Texas
  - Consultants in Cardiology, Fort Worth, Texas
  - University of Texas Division of Cardiology, Galveston, Texas
  - Methodist DeBakery Heart Center Cardiovascular Imaging Institute, Houston, Texas
  - University of Texas Health Science Center Memorial Hermann Heart & Vascular Institute, Houston, Texas
  - Harborview Medical Center Department of Cardiology, Seattle, Washington
  - Heart Clinics Northwest, Spokane, Washington
  - Inland Cardiology, Spokane, Washington
  - Northwest Cardiovascular Research Institute Spokane Cardiology, Spokane, Washington